CLINICAL TRIAL: NCT00616473
Title: The Impact of Quality End-of-Life Care in Nursing Homes
Brief Title: Quality End-of-Life Care in Nursing Homes
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0433-06-FB; 7R01NR009547-02 (NIH)
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Quality of End-of-life Care in Nursing Homes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1 Nursing Home Staff: Direct care staff
- 2 Family Members: Family members/Significant other of nursing home resident.

SUMMARY:
The purpose of this study is to examine key organizational structures and processes (leadership, teamwork, communication, palliative care) and their impact on the quality of end-of-life care for dying residents and their family members.

DETAILED DESCRIPTION:
As the American population ages, nursing homes are rapidly becoming a dominant site for death. Currently, 25% of all deaths occur in nursing homes and 35% of all elders over the age of 85 die in nursing homes. By 2020, 40% of those over 65 will die in nursing homes. Nursing home residents die in pain with undue psychosocial suffering. For all permanently placed residents, death is inevitable. Nonetheless, how residents die, is not.

There have been long standing concerns about the quality of care and quality of life in nursing homes. Although there is some evidence that the quality of care for nursing home residents has improved, serious problems continue in areas that potentially affect end-of-life such as dehydration, pressure ulcers, and pain. Efforts to improve care have rarely considered the dynamic nature of nursing home structure and process factors, such as staffing levels, leadership of the director of nursing, or communication and teamwork among staff that facilitate or impede the organization's ability to improve care processes. Findings from our preliminary studies in nursing homes indicate that organizational structure and process factors make a difference in end-of-life care for residents and their family members. More specifically, staff education, staffing levels, leadership of the Director of Nursing (DON) and administrator, teamwork and communication among direct care staff, and incorporating palliative care clinical practices into day-to-day care had a profound impact on outcomes such as the honoring of end-of-life preferences, symptom management, and satisfaction with care. A more generalizable understanding of key structure and process factors and their relationship to resident care and outcomes at the end-of-life will provide a foundation for future intervention studies aimed at improving care.

ELIGIBILITY:
Inclusion Criteria (Nursing Homes):

* 60 beds or greater

Exclusion Criteria (Nursing Homes):

* less than 60 beds

Inclusion Criteria (Nursing Home Staff):

* 19 years of age or older
* trained to provide resident care

Exclusion Criteria (Nursing Homes):

* less than 19 years of age
* staff on units exclusively Medicare or average length of stay less than 30 days

Inclusion Criteria (Family Member/Significant Other):

* 19 years of age or older
* somewhat to very involved in resident's care and decision-making

Exclusion Criteria (Family Member/Significant Other):

* not involved in resident's care and decision-making
* resident was in the nursing home less than 31 days
* resident was less than 65 years old

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nursing Homes in Nebraska and the Western half of Iowa, nursing home staff, and family members/significant other of nursing home residents
Sampling Method: Non-Probability Sample
Enrollment: 7169 (Actual)
Dates: Start 2006-12-15 (Actual); Primary Completion 2011-01-01 (Actual); Study Completion 2011-01-01 (Actual)

PRIMARY OUTCOMES:
Palliative care influence | At beginning of study (baseline), then again after 25 nursing home residents have died (assessed for 7 years)
  Questionnaires (nursing home staff and family members) to assess the influence of palliative care on staff performance (communication, leadership, and teamwork).

SECONDARY OUTCOMES:
Staffing and quality of end-of-life care | At beginning of study (baseline), then again after 25 nursing home residents have died (assessed for 7 years)
  Questionnaires (nursing home staff and family members) to assess the associations among structure (staffing), non-clinical (communication, leadership, teamwork) and clinical (palliative care) care processes and quality of end-of-life care.
Modelling nursing home palliative care | At beginning of study (baseline), then again after 25 nursing home residents have died (assessed for 7 years)
  Questionnaires (nursing home staff and family members) to assess modelling of nursing home palliative care (Unruh and Wan's expanded structure, process, and outcomes model).

CONTACTS AND LOCATIONS:
Overall Officials: Sarah A Thompson, RN, PhD, Principal Investigator — University of Nebraska; Virginia Tilden, RN, DNSC, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States